CLINICAL TRIAL: NCT03971604
Title: The Correlation Between Vitamin A / E Levels and Preeclampsia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: W2016CWZJ07
Record Dates: First submitted 2019-05-14; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Preeclampsia; Vitamin A Deficiency; Vitamin E Deficiency
MeSH Terms: conditions — Pre-Eclampsia; Vitamin A Deficiency; Vitamin E Deficiency | interventions — Vitamin A; Vitamin E

STUDY DESIGN:
Intervention Model Description: Group 1: Treated with VA, Group 2: Treated with VE, Group 3: Treated with VA+VE. To evaluate and compare the blood pressure, weight, uterine height, abdominal circumference, fetal b-mode ultrasound, blood results (blood routine, including blood VA/VE level), methods of termination of pregnancy, obstetric complications and neonatal conditions (including body length, weight, Apgar score, umbilical cord blood VA, VE level, etc.) among the three groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Experimental): treated with VA
  Interventions: Drug: Vitamin A
- group 2 (Experimental): treated with VE
  Interventions: Drug: Vitamin E
- group 3 (Experimental): treated with VA+VE
  Interventions: Drug: Vitamin A; Drug: Vitamin E
- group 4 (No Intervention): No intervention

INTERVENTIONS:
Drug: Vitamin A — treated with Vitamin A
  Arms: group 1; group 3
Drug: Vitamin E — treated with Vitamin E
  Arms: group 2; group 3

SUMMARY:
Vitamin A (VA) and vitamin E (VE) are fat-soluble vitamins and indispensable substances in life activities.

VA plays an important role in visual function, normal formation and development of epithelial cells, development and growth of bones, immune function and reproductive health. VA is of great significancCe for the growth and development of embryonic cells, especially for the development of fetal vertebrae, spinal cord, limbs, heart, eyes and ears. The lack of maternal VA will lead to the stunted development of fetal organs and tissues, and even fetal developmental malformation. In addition, VA has a protective effect on neonatal lung maturation.VA deficiency can cause the decrease in the activity of enzymes needed to catalyze the formation of progesterone precursors in pregnant women, reduce the production of steroids in adrenal glands, gonads and placenta, and seriously affect the functions of multiple organs such as heart, liver and skeletal muscle in pregnant women.

VE, also known as tocopherol, has non-enzymatic antioxidant function, and maintains the balance of REDOX reaction in vivo by efficiently removing free radicals generated by lipid peroxidation.VE can increase the synthesis of nitric oxide (NO) in endothelial cells and improve vascular endothelial function. Long-term administration of VE can improve the impaired endothelium-dependent vasodilatory function in patients.VE can promote sex hormone secretion, improve fertility and prevent abortion. Pregnancy women the body's metabolism, increases produce free radicals, lipid peroxidation, low levels of VE will result in the accumulation of excess free radicals, cause the placenta aging, vascular endothelial damage, increase the risk of the occurrence of PHI and adverse outcome rate, as well as the membranes of cell membrane damage, increase the risk of premature rupture of membranes.

Gestational hypertension is a group of diseases with both pregnancy and elevated blood pressure, and is the main cause of increased maternal and perinatal mortality, mainly including gestational hypertension, preeclampsia PE, and eclampsia, as well as chronic hypertension with preeclampsia and chronic hypertension with pregnancy. The cause of PE is unknown, but studies have found that it may be related to insufficient recast of spiral uterine arterioles, excessive activation of inflammatory immune system, damage of vascular endothelial cells, genetic factors, nutritional deficiency and insulin resistance. Recent studies have found that free radical oxidative damage may also be one of the main reasons for the occurrence and development of PE. PE occurs, the placenta bed vasospasm, ischemia, angiogenesis blocking and endothelial atherosclerotic changes, local immune cell activity, make produce free radicals increases, interfere with the vascular endothelial cell function, reduce vascular relaxation material synthesis, and shrink blood vessels increase material synthesis, promote vascular spasm, platelet condensed state is changed, thus appeared a series of PE.

Previous studies have shown that oxygen free radicals and lipid peroxides are increased in PHI patients, while the levels of VA and VE are closely related to the antioxidant capacity of the body, and their lack can lead to the imbalance of the homeostasis of redox reaction in multi-tissue cells in the body. Since both VA and VE belong to fat-soluble vitamins and are widely distributed in daily food, whether their effects on the occurrence and development of PE are independent or combined will be a question for us to explore. Therefore, this study intends to evaluate the correlation between VA, VE and VA+VE and PE occurrence through multi-center clinical studies, and explore and summarize the feasibility of VA and VE in PE adjuvant treatment.

DETAILED DESCRIPTION:
Vitamin A (VA) and vitamin E (VE) are fat-soluble vitamins, which participate in the metabolism of important substances in the body and are indispensable substances in life activities.

VA, also known as retinol, plays an important role in visual function, normal formation and development of epithelial cells, development and growth of bones, immune function and reproductive health. During fetal development, VA affects cell differentiation and proliferation by regulating gene expression, which is of great significance for the growth and development of embryonic cells, especially for the development of fetal vertebrae, spinal cord, limbs, heart, eyes and ears. Maternal lack of VA will lead to the fetal,s organ tissue dysplasia, even serious fetal development deformity. In addition, VA can promote the growth of columnar epithelial cells on the surface of alveoli, and has a certain protective effect on the maturation of neonatal lungs. VA deficiency can cause the decrease in the activity of enzymes needed to catalyze the formation of progesterone precursors in pregnant women, reduce the production of steroids in adrenal glands, gonads and placenta, and seriously affect the functions of multiple organs such as heart, liver and skeletal muscle in pregnant women.

VE, also known as tocopherol, has non-enzymatic antioxidant function, and maintains the balance of REDOX reaction in vivo by efficiently removing free radicals generated by lipid peroxidation.VE can increase the synthesis of nitric oxide (NO) in endothelial cells, release electrons to stabilize free radicals, protect NO from inactivation of free radicals, and improve vascular endothelial function. Long-term use of VE has been found to improve endothelium-dependent vasodilation in patients with impaired vasodilation.VE can promote sex hormone secretion, improve fertility, prevent abortion, clinically commonly used VE treatment threatened abortion and habitual abortion. Pregnancy women the body's metabolism, increases produce free radicals, lipid peroxidation, low levels of VE will result in the accumulation of excess free radicals, which cause the placenta aging, vascular endothelial damage, increase the risk of the occurrence of PIH and adverse outcome rate, and cell membrane damage of membranes, the occurrence of premature rupture of membranes increased risk.

Gestational hypertension disease is a group of disease and high blood pressure, pregnancy rate is about 5% - 12%, serious impact on maternal and child health, is a major cause of maternal and perinatal mortality increase, mainly including gestational hypertension, preeclampsia preeclampsia (PE), eclampsia, and chronic hypertension complicated by preeclampsia and chronic hypertension with pregnancy. Preeclampsia is the most common type, including mild and severe preeclampsia, of which severe preeclampsia accounts for about 30% to 50%.The cause of PE is unknown, but studies have found that it may be related to insufficient recast of spiral uterine arterioles, excessive activation of inflammatory immune system, damage of vascular endothelial cells, genetic factors, nutritional deficiency and insulin resistance. Recent studies have found that free radical oxidative damage may also be one of the main reasons for the occurrence and development of PE.PE occurs, the placenta bed vasospasm, ischemia, angiogenesis blocking and endothelial atherosclerotic changes, strengthen local immune cell activity, increase the free, free radical and lipid peroxide interfere with the vascular endothelial cell function, make blood-vessel loose material such as nitric oxide (NO), top ring element synthesis reduce I2, materials and shrink blood vessels, such as endothelin (ET), thromboxane A2, such as synthetic increase, promote vascular spasm, platelet condensed state is changed, thus appeared a series of PE.

Previous studies have shown that oxygen free radicals and lipid peroxides increase in the body of patients with PIH, and excessive antioxidants are consumed. However, the levels of VA and VE are closely related to the antioxidant capacity of the body, and the lack of them can lead to the imbalance of redox reaction homeostasis in multi-tissue cells in the body, thus resulting in the occurrence of oxidative stress in the body. Studies have found that oxidative stress can cause the occurrence and development of PE when the levels of VA and VE are reduced. Therefore, it is not clear whether the application of VA and VE can reduce the incidence of PE and improve the prognosis of neonates. Since both VA and VE belong to the family of fat-soluble vitamins and are widely present in daily food, are they independent or combined in influencing the occurrence and development of PE. Therefore, this study intends to evaluate the correlation between VA, VE and VA+VE in PE during pregnancy through multi-center clinical studies, and explore and summarize the feasibility of VA and VE in PE adjuvant treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years of natural pregnancy, early pregnancy without threatened abortion and infection
2. No history of hypertension, diabetes, heart disease and other internal and surgical diseases
3. Pregnancy are normal to take folic acid and calcium tablets, did not take other drugs
4. Agree to participate in the experiment and sign the informed consent

Exclusion Criteria:

1. Refuse to sign or request to withdraw the informed consent midway
2. Serious adverse events, allergies or intolerance
3. Poor patient compliance, refused to cooperate with the experimental requirements

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
To compare the serum VA and VE levels between normal pregnant women and pre-eclampsia pregnant women | change from 20 to 37 weeks
  To compare the serum VA and VE levels between normal pregnant women and pre-eclampsia pregnant women
To compare the levels of VA and VE in pregnant women with mild and severe preeclampsia | change from 20 to 37 weeks
  To compare the levels of VA and VE in pregnant women with mild and severe preeclampsia
To analyze the changes in serum levels of VA and VE in pregnant women with mild and severe preeclampsia, as well as the effects of independent and combined intake of VA and VE on the disease | change from 20 to 37 weeks
  To analyze the changes in serum levels of VA and VE in pregnant women with mild and severe preeclampsia, as well as the effects of independent and combined intake of VA and VE on the disease
To analyze the correlation between serum VA and VE levels in the case group and important indicators related to the disease (such as blood pressure, body weight, hematuria routine, liver and kidney function, etc.) . | change from 20 to 37 weeks
  To analyze the correlation between serum VA and VE levels in the case group and important indicators related to the disease (such as blood pressure, body weight, hematuria routine, liver and kidney function, etc.) .

CONTACTS AND LOCATIONS:
Overall Officials: liquan wang, Study Director — 2th affiliated hospital of medical college of zhejiang university
Locations (1):
- The second affiliated hospital of medical college of zhejiang university, Hangzhou, Zhejiang, China